CLINICAL TRIAL: NCT06045377
Title: Effect of a Nutraceutical, Containing Red Yeast Rice and Polycosanols (Armolipid), on Lipid Profile in Children With Moderate and Severe Hypercholesterolemia.
Brief Title: Effect of Armolipid on Lipid Profile in Children With Hypercholesterolemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Athens General Children's Hospital "Pan. & Aglaia Kyriakou" (Other)
Responsible Party: Principal Investigator, Achilleas Attilakos, Assoc. Prof. of Pediatrics, Athens General Children's Hospital "Pan. & Aglaia Kyriakou"
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1474/10 Jan 2020
Record Dates: First submitted 2023-08-29; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Dyslipidemias; Children, Only
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Armolipid (Experimental): One tablet of Armolipid (Rottapharm S.p.A., Monza, Italia), containing 200 mg red yeast rice, 10 mg policosanols, 0.2 mg folic acid, 2.0 mg coenzyme Q10 and 0.5 mg astaxanthin was administered once-daily with lunch.
  Clinical and laboratory evaluation took place before and 6 (IQR: 5-8) and 16 (IQR: 11-19.7) months after treatment.
  Interventions: Dietary Supplement: Effect of Armolipid on Lipid Profile in Children With Hypercholesterolemia

INTERVENTIONS:
Dietary Supplement: Effect of Armolipid on Lipid Profile in Children With Hypercholesterolemia — A prospective single center cohort study

SUMMARY:
Data concerning the effectiveness od nutraceuticals in children with dyslipidemia are lacking. The aim of the present study was to evaluate the efficacy and safety of the long-term use of a dietary supplement containing red yeast rice (RYR), combined with other natural compounds, in children and adolescents with hypercholesterolemia.

A nutraceutical, containing RYR, polycosanols, coenzyme Q10, astaxanthin and folic acid (commercial name: Armolipid), was administered once-daily in 84 children/adolescents with moderate or severe hypercholesterolemia.

DETAILED DESCRIPTION:
This is a prospective single center cohort study conducted at Outpatient Lipid Unit of 2nd Department of Pediatrics of the National and Kapodistrian University of Athens at the "Panagiotis & Aglaia Kyriakou" Children's Hospital in Greece. The study complies with the Declaration of Helsinki and the protocol was reviewed and approved by the appropriate ethical committee. Parental informed written consent was obtained prior to enrollment.

Study population: Ninety children and adolescents, aged 7 to 16 years, with primary dyslipidemia.

All participants had a positive family history for hypercholesterolemia (LDL > 95th percentile) and most of them had a positive family history for premature CVD (<55 years for males and <60 years for females) in first or/and second-degree relatives. Eleven of them had a genetically confirmed diagnosis of HeFH, while the rest had a probable or positive HeFH according to the Dutch Lipid Clinic Network criteria. None of them had moderate or significant hypertriglyceridemia, even those with increased body mass index (BMI).

All children followed a low saturated fat and low cholesterol diet by a trained dietician and had moderate or intense physical activity, for at least 6 months before the participation in the study. In addition, during the last 6 months, 19 of them consumed 1.5 - 2.5g of plant sterols daily in the form of a yogurt drink or spread. Lifestyle and eating habits were maintained throughout the study.

A nutraceutical containing five natural substances formulated as a tablet with the commercial name Armolipid (Rottapharm S.p.A., Monza, Italia), was recommended in all participants. Every tablet contained 200 mg red yeast rice (RYR) extract equivalent to 3 mg of monacolin K, 10 mg policosanols, 0.2 mg folic acid, 2.0 mg coenzyme Q10 and 0.5 mg astaxanthin, and was citrinin-free. It was administered once-daily with lunch.

All participants as well as their parents were interviewed using a data collection form, created specifically for this research. Details concerning compliance to supplement intake, as well as possible adverse effects were recorded and analysed. Six out of 90 children were excluded from the study because they did not comply with the recommendation for taking the supplement (compliance rate 93.3%). All the rest 84 children had one and 64 of them had two evaluations under Armolipid treatment.

Clinical and Labolatory evaluation: A clinical and laboratory evaluation of all participants took place right before (Time 0, T0) and once (n=84, Time 1, T1) or twice (n=64, T1 and Time 2, T2) after the start of nutraceutical supplementation.

The body weight (BW) in kg, the height (H) in cm were measured to the nearest 0.1 kg and 0.5 cm, respectively (TANITA, Corporation Tokyo), with children barefoot and lightly dressed. BMI was calculated as BW in kg per H in m2. The standard deviation scores (z-scores) of BW, H and BMI were also calculated according to a standardized age- and sex- specific calculator. Waist circumference (WC) in cm was measured and the ratio of WC/Height was calculated. Systolic (SBP) and diastolic blood pressure (DBP) in mmHg were measured three consecutive times using an automated oscillometric device (Dinamap V100, GE Medical Systems Information Technologies) and the average value of the three measurements was used in the statistical analysis. The stage of puberty was recorded according to Tanner stages (I-V) for boys and girls.

A full lipid profile including TC, LDL-C, high density lipoprotein - cholesterol (HDL-C), non-high density lipoprotein - cholesterol (non-HDL-C), triglycerides (TGs), apolipoprotein A1 (Apo-A1), apolipoprotein B (Apo-B), and lipoprotein (a) [Lp(a)] levels was evaluated in serum, after an overnight fast. Serum creatinine, glucose, aspartate and alanine aminotransferases (AST and ALT), creatine kinase (CK), and thyroid-stimulating hormone (TSH) were also assessed. A full blood count was performed in all participants.

TC, HDL-C, LDL-C, TGs, glucose, ALT, AST, CK and creatinine were measured using an enzymatic method (Roche Diagnostics) on an automatic analyzer (Cobass Integra 800), and Apo-A1, Apo-B, and Lp(a) by an immunonephelometric assay (Siemens BNII Nephelometer Analyzer), with an intra-assay and inter-assay variation <5% for all tests. Non-HDL-C was measured as TC minus HDL-C. All lipid values are expressed in mg/dL. Haematological parameters (full blood count) were analyzed using the SysmexXE-2100 automated haematology analyzer (Roche Diagnostics). All tests were performed according to the manufacturers' instructions.

At the time of the examination, all children were healthy and none of them had a febrile or afebrile infection in the two weeks preceding the check-up.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C >150 mg/dl in more than two measurements, after therapeutic lifestyle changes for at least 6 months.

Exclusion Criteria:

* Secondary hypercholesterolemia
* Presence of any chronic disease or growth and developmental disorders
* Abnormal liver, kidney or thyroid function
* Prior use of hypolipidemic or other medication, at least 6 months before participation in the study.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Levels of LDL-C serum levels | Laboratory evaluation before and 6 and 16 months after treatment
  LDL-C levels were evaluated in serum, after an overnight fast.

SECONDARY OUTCOMES:
Improvement of other than LDL-C parameters of lipid profile, as well as the evaluation of hepatic and muscle enzymes elevation. | Laboratory evaluation before and 6 and 16 months after treatment
  A lipid profile including TC, high density lipoprotein - cholesterol (HDL-C), non-high density lipoprotein - cholesterol (non-HDL-C), triglycerides (TGs), apolipoprotein A1 (Apo-A1), apolipoprotein B (Apo-B), and lipoprotein (a) [Lp(a)] levels was evaluated in serum, after an overnight fast. Serum creatinine, aspartate and alanine aminotransferases (AST and ALT) and creatine kinase (CK) were also assessed.

OTHER OUTCOMES:
Waist Circumference (WC) and the ratio of WC/Height | Clinical evaluation before and 6 and 16 months after treatment
  WC in cm was measured and the ratio of WC/Height was calculated.
Systolic (SBP) and diastolic blood pressure (DBP) | Clinical evaluation before and 6 and 16 months after treatment
  SBP and DBP in mmHg were measured three consecutive times using an automated oscillometric device (Dinamap V100, GE Medical Systems Information Technologies).
Body weight in kg | Clinical evaluation before and 6 and 16 months after treatment
  The body weight (BW) in kg, measured to the nearest 0.1 kg (TANITA, Corporation Tokyo), with children barefoot and lightly dressed.
Body height in cm | Clinical evaluation before and 6 and 16 months after treatment
  The body height (H) in cm, measured to the nearest 0.5 cm, (TANITA, Corporation Tokyo), with children barefoot.
BMI (calculated as body weight in kg per height in m2) | Clinical evaluation before and 6 and 16 months after treatment
  BMI was calculated as BW in kg per H in m2. The standard deviation scores (z-scores) of BW, H and BMI were also calculated according to a standardized age- and sex- specific calculator.

CONTACTS AND LOCATIONS:
Overall Officials: Achilleas Attilakos, Assoc.Prof, Principal Investigator — Athens Children's Hospital Pan. and Aglaia Kyriakou
Locations (1):
- Lipid Outpatient Unit, 2nd Department of Pediatrics, Medical School, National and Kapodistrian University of Athens (NKUA), "P. & A. Kyriakou" Children's Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watts GF, Gidding SS, Hegele RA, Raal FJ, Sturm AC, Jones LK, Sarkies MN, Al-Rasadi K, Blom DJ, Daccord M, de Ferranti SD, Folco E, Libby P, Mata P, Nawawi HM, Ramaswami U, Ray KK, Stefanutti C, Yamashita S, Pang J, Thompson GR, Santos RD. International Atherosclerosis Society guidance for implementing best practice in the care of familial hypercholesterolaemia. Nat Rev Cardiol. 2023 Dec;20(12):845-869. doi: 10.1038/s41569-023-00892-0. Epub 2023 Jun 15. PMID 37322181
- [Background] Santini A, Novellino E. Nutraceuticals in hypercholesterolaemia: an overview. Br J Pharmacol. 2017 Jun;174(11):1450-1463. doi: 10.1111/bph.13636. Epub 2016 Oct 29. PMID 27685833
- [Background] Cicero AFG, Fogacci F, Stoian AP, Vrablik M, Al Rasadi K, Banach M, Toth PP, Rizzo M. Nutraceuticals in the Management of Dyslipidemia: Which, When, and for Whom? Could Nutraceuticals Help Low-Risk Individuals with Non-optimal Lipid Levels? Curr Atheroscler Rep. 2021 Aug 4;23(10):57. doi: 10.1007/s11883-021-00955-y. PMID 34345932
- [Background] Cicero AFG, Kennedy C, Knezevic T, Bove M, Georges CMG, Satrauskiene A, Toth PP, Fogacci F. Efficacy and Safety of Armolipid Plus(R): An Updated PRISMA Compliant Systematic Review and Meta-Analysis of Randomized Controlled Clinical Trials. Nutrients. 2021 Feb 16;13(2):638. doi: 10.3390/nu13020638. PMID 33669333
- [Background] Guardamagna O, Abello F, Baracco V, Stasiowska B, Martino F. The treatment of hypercholesterolemic children: efficacy and safety of a combination of red yeast rice extract and policosanols. Nutr Metab Cardiovasc Dis. 2011 Jun;21(6):424-9. doi: 10.1016/j.numecd.2009.10.015. Epub 2010 Feb 12. PMID 20153154